CLINICAL TRIAL: NCT00705172
Title: Efficacy and Safety of Norditropin® (Somatropin) in Children With Prader-Willi Syndrome (PWS)
Brief Title: Retrospective Observational Study on Efficacy and Safety of Norditropin® in Children With Prader-Willi Syndrome
Status: Completed | Type: Observational
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: GHLIQUID-1961
Record Dates: First submitted 2008-06-24; First posted 2008-06-25 (Estimated); Last update posted 2023-11-02 (Actual); Status verified 2023-10

CONDITIONS: Genetic Disorder; Prader-Willi Syndrome
MeSH Terms: conditions — Genetic Diseases, Inborn; Prader-Willi Syndrome | interventions — Human Growth Hormone

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- A
  Interventions: Drug: somatropin

INTERVENTIONS:
Drug: somatropin — Prader-Willi syndrome children treated with at least one dose of Norditropin®
  Other Names: Norditropin®

SUMMARY:
This study is conducted in Europe. The aim of this observational study is to collect data from children with Prader-Willi Syndrome, who have been treated off-label with Norditropin® for more than 12 months to seek approval for Norditropin® treatment with Prader-Willi Syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent obtained before any trial-related activities
* Genetically diagnosed Prader-Willi Syndrome
* Received at least one dose of Norditropin® treatment
* Pre-pubertal at start of treatment; assessed by Tanner stage 1, or testicular volume below 4ml (according to Tanner 1976)

Exclusion Criteria:

* Pre-treatment with other Growth Hormone preparation prior to treatment with Norditropin®

Max Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children with Prader-Willi Syndrome
Sampling Method: Non-Probability Sample
Enrollment: 41 (Actual)
Dates: Start 2008-11; Primary Completion 2008-11 (Actual); Study Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
Primary objective is to investigate changes in height Standard Deviation Score (SDS) | in response to 12 months Norditropin® treatment in children with PWS (referenced to PWS population

SECONDARY OUTCOMES:
Changes in height SDS from start of treatment to last observation during Norditropin treatment (referenced to PWS population1) | at 12 months- and at last observation during Norditropin treatment
Change in body composition (DEXA, Bio impedance or stable isotope dilution) | at 12 months- and at last observation during Norditropin treatment
Height velocity (HV) and change in HV | at 12 months- and at last observation during Norditropin treatment
Glycated Fraction of Haemoglobin (HbA1c) | at 12 months- and at last observation during Norditropin treatment
Insulin-Like Growth Factor-I (IGF-I) | at 12 months- and at last observation during Norditropin treatment
Haematology | at 12 months- and at last observation during Norditropin treatment
Thyroid-stimulating hormone (TSH) and active form of free thyroxin | at 12 months- and at last observation during Norditropin treatment
Adverse Events. | at 12 months- and at last observation during Norditropin treatment

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (3):
- Arhus N, Denmark
- Hildesheim, Germany
- Zurich, Switzerland

REFERENCES:
- [Derived] Meinhardt U, Christiansen JS, Farholt S, Lammer C, Ostergaard JR, Schmidt F, Kappelgaard AM, Eiholzer U. The efficacy and safety of long-term Norditropin(R) treatment in children with Prader-Willi syndrome. Horm Metab Res. 2013 Jul;45(7):532-6. doi: 10.1055/s-0033-1343449. Epub 2013 Apr 30. PMID 23632904
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com